CLINICAL TRIAL: NCT03698045
Title: Study to Evaluate the Safety and Tolerability of Pro-143 Ophthalmic Solution in Healthy Volunteers.
Brief Title: Safety and Tolerability of PRO-143 Ophthalmic Solution in Healthy Volunteers.
Acronym: PRO-143
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: the clinical study was canceled by the sponsor due to logistics and programming
Sponsor: Laboratorios Sophia S.A de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOPH143-0212/I; PRO-143
Record Dates: First submitted 2012-02-22; First posted 2018-10-05 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Conjunctivitis, Bacterial
Keywords: PRO-143; Topical antibiotic; Ophthalmic antibiotic; External bacterial infections
MeSH Terms: conditions — Conjunctivitis, Bacterial | interventions — apolipoprotein A-I Giessen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PRO-143 Ophthalmic Solution (Experimental): PRO-143 Ophthalmic Solution applied four times per day (c/6 hours) during 10 days.
  Interventions: Drug: PRO-143 Ophthalmic Solution

INTERVENTIONS:
Drug: PRO-143 Ophthalmic Solution — PRO-143 Ophthalmic Solution applied four times per day (C/6 hours) during 10 days.
  Other Names: PRO-143

SUMMARY:
Study to evaluate the safety and tolerability of PRO-143 solution ophthalmic in healthy volunteers.

DETAILED DESCRIPTION:
A phase I, open label and unicentric clinical trial to evaluate the safety and tolerability of PRO-143 ophthalmic solution in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female.
* Age ≥ 18 years old at screening visit.

Exclusion Criteria:

* Any ocular or systemic condition.
* Patient with one blind eye.
* Visual acuity of 20/40 in any eye.
* Use of ocular or systemics medications.
* Contraindications or sensitivity to any component of the study treatments.
* Contact lens users.
* Ocular surgery within the past 3 months..
* Women who were not using an effective means of contraception or who were pregnant or nursing.
* Participation in any studies of investigational drugs within 90 days previous to the inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-11; Primary Completion 2014-02 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Conjunctival bulbar hyperemia | 10 days
  Conjunctival hyperemia is defined as the simplest reaction of the conjunctiva to a stimulus, a red appearance secondary to the vasodilation of the conjunctival vessels of variable intensity. He will graduate using the Efron scale.
  0 Normal , 1 Very slight, 2 Mild, 3 Moderate, 4 Severe.
Number of Participants with adverse events | 10 days
  he evaluation of adverse events requires a questioning conducted by the principal investigator and the appropriate exploratory techniques for its detection. the number of adverse events per study group will be considered for the analysis

SECONDARY OUTCOMES:
Intraocular pressure (IOP) | 10 days
  Tonometry is the objective measure of Intraocular pressure, based primarily on the force required to flatten the cornea, or the degree of corneal indentation produced by a fixed force. Goldman's tonometry is based on the Imbert-Fick principle. the result will be expressed in millimeters of mercury and the comparison between groups will be carried out.
Visual ability (VA) | 10 days
  The VA will be evaluated basally, without refractive correction with the Snellen chart. Which will be located in a place with adequate lighting, natural or artificial and at a distance of 3 meters from the subject to be evaluated
Eye comfort index (ICO) | 10 days
  It is a questionnaire designed to measure the irritation of the ocular surface with Rasch analysis to produce estimates on a linear scale of intervals (ratings: 0-100). Similar to the index for ocular surface diseases, the ocular comfort index (ICO) evaluates symptoms. The ICO contains 6 items that focus on the discomfort associated with the ocular surface. Each of these questions has two parts, which inquire separately the frequency and severity of the symptoms.
  The evaluator will deliver the questionnaire to the subject and allow the subject to answer it calmly without any pressure and / or coercion, will only assist him if he has difficulty understanding any of the questions.

CONTACTS AND LOCATIONS:
Overall Officials: José F Alaniz-De La O, MD, Principal Investigator — Independent Clinical Research Center; Laura R Saucedo-Rodíguez, MD, Principal Investigator — Independent Clinical Research Center; Leopoldo M Baiza-Durán, MD, Study Director — Clinical Research Department. Laboratorios Sophia SA de CV
Locations (1):
- Independent Clinical Research Center, Guadalajara, Jalisco, Mexico